CLINICAL TRIAL: NCT04399824
Title: Focal Radiation Therapy (FRaT) Trial in Patients With Low/Intermediate-Risk Prostate Cancer
Brief Title: Focal Radiation Therapy for the Treatment of Low or Intermediate-Risk Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not open
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-000051; NCI-2020-01464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-000051 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-03-24; First posted 2020-05-22 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (SBRT) (Experimental): Patients undergo SBRT in 5 fractions over 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Arm II (HDR brachytherapy) (Experimental): Patients undergo HDR brachytherapy on day 1 and a second fraction within 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: High-Dose Rate Brachytherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy — Undergo HDR brachytherapy
  Other Names: Brachytherapy, High Dose
  Arms: Arm II (HDR brachytherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm I (SBRT)

SUMMARY:
This phase II trial studies how well focal radiation therapy with stereotactic body radiation therapy (SBRT) or high-dose rate (HDR) brachytherapy works in treating patients with low or intermediate-risk prostate cancer. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Brachytherapy, also known as internal radiation therapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. HDR brachytherapy uses high doses of radiation to target these tumor cells. Giving focal radiation therapy with SBRT or HDR brachytherapy may target dominant tumor cells while sparing the reminder of the prostate or surrounding normal organs and ultimately reduce side effects while maintaining disease control.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate biochemical progression free survival (bPFS) using the Phoenix definition.

II. Changes in quality of life. IIa. Prostate-Quality of Life (PR-QOL). IIb. Expanded Prostate Cancer Index Composite (EPIC).

SECONDARY OBJECTIVES:

I. Prostate-specific antigen (PSA) response at 3, 6, 12, and 24 months. II. Clinical progression free survival. IIa. Including phoenix definition, local progression by Response Evaluation Criteria in Solid Tumors (RECIST), regional progression, distant metastasis, or death.

III. Distant metastasis free survival. IV. Development of castration-resistant disease. V. Overall survival.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients undergo SBRT in 5 fractions over 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo HDR brachytherapy on day 1 and a second fraction within 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 weeks, every 3 months for up to 24 months, every 6 months for up to 60 months, and then every 8-12 months until 120 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma within 90 days prior to registration via systematic biopsy and with the following low/intermediate-risk features:

  * cT1c - T2b
  * PSA =< 15
  * < 50% cores positive
  * Gleason score (GS) =< 7 (3+4 and 4+3 included)
* Multiparametric magnetic resonance imaging (MRI) (mp-MRI) confirmed lesion(s) with only one lobe involvement of the prostate
* Unilateral disease on systematic biopsy
* No distant or locally advanced disease on standard staging exams as indicated

  * Bone scan and abdominopelvic computed tomography (CT)/MRI OR
  * Prostate specific membrane antigen (PSMA) positron emission tomography (PET)
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status 0/1 within 60 days prior to enrollment

Exclusion Criteria:

* Gleason score >= 8
* Gross extracapsular extension
* Seminal vesicle invasion
* Radiographic nodal or distant metastatic disease
* Androgen deprivation therapy within 90 days of enrollment
* Lesion(s) comprising > 40% of total prostate volume
* Lesion < 0.5 cm from urethra
* Prior radical prostatectomy
* Prior radiotherapy to the pelvis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Biochemical progression free survival | At 5 years
  Will be assessed using the Phoenix definition and obtained via Kaplan-Meier analysis to provide an overview of efficacy for focal radiation therapy.
Incidence of adverse events | Up to 120 months (10 years)
  Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0. Will be defined as the percentage of patients who encounter adverse events and calculated to indicate the toxicity level of focal radiation therapy.
Change in quality of life | Baseline up to 120 months
  Will be assessed using Prostate-Quality of Life and Expanded Prostate Cancer Index Composite. The change of the two scores will be assessed via two-sided paired t-test.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) response | At 3, 6, 12, and 24 months
  PSA response of each patient at 3, 6, 12, and 24 months will be collected and the PSA changes from baseline PSA to each time point will be evaluated via two-sided paired t-test.
Clinical progression free survival | At 5 years
Distant metastasis free survival | At 5 years
  Will be obtained via Kaplan-Meier analysis to provide an overview of efficacy for focal radiation therapy.
Development of castration-resistant disease | Up to 120 months (10 years)
  Defined as clinical/biochemical progression of prostate cancer with testosterone <40 ng/dl [nanograms (ng) per deciliter (dL)]
Overall survival | At 5 years
  Will be obtained via Kaplan-Meier analysis to provide an overview of efficacy for focal radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Lee, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States